CLINICAL TRIAL: NCT03240302
Title: A Comparative Study of Sibling Oocytes, Which Examines Two Sperm Selection Methods for Top Quality of Spermatozoa , Prior Intracytoplasmic Sperm Injection (ICSI) Performance, and Their Effect on Embryo Quality and IVF Outcome: A Common Selection Method Based on Morphology (ICSI) vs. a Selection Method for Mature Spermatozoa With CD44 Receptors for Hyaluronic Acid (PICSI - Physiological Selected Intracytoplasmic Sperm Injection)
Brief Title: A Comparative Study of Sibling Oocytes: ICSI vs. the PICSI Sperm Selection Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-0069-17
Record Dates: First submitted 2017-07-31; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSI Procedure (Active Comparator): The ICSI procedure is the standard procedure of selection and injection of sperm into the oocyte using a standard ICSI petri dish.
  Interventions: Device: ICSI petri dish
- PICSI Procedure (Active Comparator): The PICSI procedure is based on a selection of mature spermatozoa with CD44 receptors and their injection into the oocyte using the PICSI petri dish that has been coated with hyaluronic acid on its bottom.
  Interventions: Device: PICSI petri dish

INTERVENTIONS:
Device: ICSI petri dish — Half of the oocytes will be placed into the standard ICSI petri dish and they will be injected with sperm with normal morphology.
  Arms: ICSI Procedure
Device: PICSI petri dish — Half of the oocytes will be placed into a PICSI petri dish (whose bottom is coated with hyaluronic acid) and the mature spermatozoa with CD44 receptors that are attached to the bottom of the dish will be injected into them.
  Arms: PICSI Procedure

SUMMARY:
The aim of this research is to compare sibling oocytes using two sperm selection methods for choosing the best quality spermatozoa before they are injected into oocytes and the influence of each of these methods on embryo quality and IVF outcome.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-60
* Females aged 18-35
* Males with mild OTA (oligo terato astheno zoospermia) and at least one failed IVF cycle
* Males with normozoospermia with at least 2 unexplained failed IVF cycles
* Females with normal FSH and normal AMH values
* Females who have retrieved in previous cycles at least 6 oocytes

Exclusion Criteria:

* Couples who have been exposed to heavy smoking, drugs and chronic diseases
* Males who have undergone testicular surgery (TESE) or defined as severe OTA
* Females with egg factor infertility

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of fertilization rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The fertilization rates of the ICSI and PICSI methods will be compared.
Comparison of embryo quality | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The embryo quality of the ICSI and PICSI methods will be compared.

SECONDARY OUTCOMES:
Implantation rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The implantation rates of the ICSI and PICSI methods will be compared.
Pregnancy rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The pregnancy rates of the ICSI and PICSI methods will be compared.
Miscarriage rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The miscarriage rates of the ICSI and PICSI methods will be compared.
Live birth rate | Three years
  Injected sibling oocytes are incubated in a time-lapse incubator which enables ongoing observation after fertilization and cleavage of each oocyte. The live birth rates of the ICSI and PICSI methods will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Einat Shalom Paz, MD, Principal Investigator — Hillel Yaffe Medical Center; Medeia Michaeli, PhD, Study Director — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No